CLINICAL TRIAL: NCT03816228
Title: Imaging of Brain Structural/Functional Connectivity and Amyloid and Tau Lesions in APOE4 Carriers. (IND 123119, Protocol Z)
Brief Title: Imaging of Brain Structural/Functional Connectivity and Amyloid and Tau Lesions in APOE4 Carriers.
Acronym: Protocol_Z
Status: Withdrawn | Type: Observational
Why Stopped: We will capture subjects under another study
Sponsor: Tammie L. S. Benzinger, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Tammie L. S. Benzinger, MD, PhD, Professor of Radiology & Neurological Surgery, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Other Study IDs: IND 123119 Protocol Z
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease
Keywords: Dementia; Taupathies; Brain Disease; Mild Cognitive Impairment; Neurodegenerative Disease
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Cognitive Dysfunction; Neurodegenerative Diseases | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental Flortaucipir: Participants will receive a single intravenous bolus injection of flortaucipir along with PET imaging.
  Interventions: Drug: F 18 T807 Flortaucipir

INTERVENTIONS:
Drug: F 18 T807 Flortaucipir — Participants will receive a single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807. For those who cannot tolerate the full exam, participants will receive single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807.
  Other Names: 18F-AV-1451

SUMMARY:
To advance current knowledge on the vascular contributions to dementia

DETAILED DESCRIPTION:
This is a multi-center study at Washington University (WASH U), University of Southern California (USC), and Huntington Medical Research Institute (HMRI).The overall goal of both the AA program and the PPG program is to advance current knowledge on the vascular contributions to dementia particularly in individuals with the major genetic risk factor for late-onset AD, i.e., apolipoprotein E-ε4 (APOE4) gene that develop early vascular dysfunction and significant cerebrovascular pathology compared to non-carriers, and establish whether the neurovasculature plays a key role in cognitive decline, and therefore is a key new therapeutic target to treat dementia in APOE4 carriers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, any race
* Age > 18 years
* Participation in one of the ongoing projects affiliated with the Knight ADRC at Washington University and referred by the MAP staff and a Washington University physician.
* Normal cognition or early-stage symptomatic AD
* Females of childbearing potential without documented history of menopause or hysterectomy who do participate must not be pregnant or breastfeeding at screening
* (negative urine β-HCG within 24 hours prior to injection), and must agree to avoid becoming pregnant. Females of childbearing potential who do not agree to use reliable contraception or refrain from sexual activity for 24 hours following administration of flortaucipir injection.
* Enrollment in DCE-MRI study
* Capacity to give informed consent and follow study procedures

Exclusion Criteria:

* Any illness preventing cooperation with testing or longitudinal participation
* Exclusion from the Knight ADRC or DIAN referring project
* Has a high risk for Torsades de Pointes or is taking medications known to prolong or may prolong QT interval (refer to study attachment "Restricted Medication List").
* MRI contraindications (e.g. electronic medical devices, severe claustrophobia, inability to lie still for long periods) that make it unsafe to participate in an MRI scan, using standard screening processes implemented by Washington University and Barnes-Jewish Hospital
* Currently pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of participants currently enrolled in ongoing projects affiliated with the Knight ADRC will be recruited. Without disclosing individual genetic risk status, 202 of these participants will include a mix of APOE4/4 (~7%), APOE3/4 (~30%), and APOE3/3 (~63%) carriers. In addition, without disclosing individual mutation status, ~40 PSEN1 carriers and non-carrier family members currently enrolled in the Dominantly Inherited Alzheimer Network (DIAN) study at Washington University will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
F 18 T807 Standard Uptake Value Ratios | 5 years
  F 18 T807 Standard Uptake Value Ratios (SUVR) will be correlated with other imaging modalities (MRI, PET amyloid imaging) and cognitive performance.

CONTACTS AND LOCATIONS:
Overall Officials: Tammie Benzinger, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
We will share the data with other researchers. They may be doing research in areas similar to this research or in other unrelated areas. These researchers may be at Washington University, at other research centers and institutions, or industry sponsors of research. We may also share the research data with large data repositories (a repository is a database of information) for broad sharing with the research community. The participant"s individual research data is placed in one of these repositories only qualified researchers, who have received prior approval from individuals that monitor the use of the data, will be able to look at this information.

REFERENCES:
- [Background] Akinyemi RO, Mukaetova-Ladinska EB, Attems J, Ihara M, Kalaria RN. Vascular risk factors and neurodegeneration in ageing related dementias: Alzheimer's disease and vascular dementia. Curr Alzheimer Res. 2013 Jul;10(6):642-53. doi: 10.2174/15672050113109990037. PMID 23627757
- [Background] Fleisher A, Grundman M, Jack CR Jr, Petersen RC, Taylor C, Kim HT, Schiller DH, Bagwell V, Sencakova D, Weiner MF, DeCarli C, DeKosky ST, van Dyck CH, Thal LJ; Alzheimer's Disease Cooperative Study. Sex, apolipoprotein E epsilon 4 status, and hippocampal volume in mild cognitive impairment. Arch Neurol. 2005 Jun;62(6):953-7. doi: 10.1001/archneur.62.6.953. PMID 15956166
- [Background] Petersen RC, Doody R, Kurz A, Mohs RC, Morris JC, Rabins PV, Ritchie K, Rossor M, Thal L, Winblad B. Current concepts in mild cognitive impairment. Arch Neurol. 2001 Dec;58(12):1985-92. doi: 10.1001/archneur.58.12.1985. PMID 11735772